CLINICAL TRIAL: NCT01568021
Title: Post Market Surveillance of OZURDEX® for Branch Retinal Vein Occlusion (BRVO) and Central Retinal Vein Occlusion (CRVO)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/RET/007
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: Single dose of dexamethasone 700 ug intravitreal implant (OZURDEX®) which may be repeated over 1 year as per standard of care in clinical practice. No intervention was administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention was administered in this study.

SUMMARY:
This multicenter observational study will assess the efficacy and tolerability of OZURDEX® in clinical practice, and will assess the time at which patients are considered for retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Macular Edema
* Prescribed OZURDEX®

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with BRVO and CRVO prescribed OZURDEX®
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Glostrup Municipality, Denmark
- Oslo, Norway
- Uppsala, Sweden

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a Post-Marketing Surveillance Study of OZURDEX®. 100 participants who received OZURDEX® as standard of care in clinical practice were enrolled in the study. Only 99 participants who had data recorded at Baseline and Follow-up were included in the analyses.
Period: Overall Study
Arm/Group | OZURDEX®
Started | 99
Completed | 83
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | OZURDEX®
Number analyzed (Participants) | 99
Age, Customized [Number; unit: participants]
  < 45 years | 1
  45 to 65 years | 24
  > 65 years | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Time to First Re-treatment
Description: Time to first re-treatment was defined as the time in days between the first administration of Ozurdex® and the following administration of Ozurdex® (re-treatment) in the study eye.
Time Frame: 1 Year
Population: All Participants with complete data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | OZURDEX®
Number analyzed (Participants) | 99
days | 157 [134 to 189]

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score
Description: BCVA was measured in the study eye using an eye chart and was reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number improvement in the number of letters read means that the vision improved.
Time Frame: Baseline, Weeks 12, 24 and 48
Population: All participants with complete data at the given time-point.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 99
letters
  Baseline | 52.8 (15.61)
  Change from Baseline at Week 12 (n= 68) | 8.5 (13.16)
  Change from Baseline at Week 24 (n= 75) | 6.9 (13.01)
  Change from Baseline at Week 48 (n= 75) | 2.5 (18.61)

3. Secondary Outcome: Change From Baseline in Central Retinal Thickness as Measured by Optical Coherence Tomography (OCT)
Description: Central Retinal Thickness was measured in the study eye using OCT, a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina to assess retinal thickness. A negative change indicated an improvement.
Time Frame: Baseline, Weeks 12, 24 and 48
Population: All participants with complete data at the given time-point.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | OZURDEX®
Number analyzed (Participants) | 99
microns
  Baseline (n- 93) | 535.2 (166.75)
  Change from Baseline at Week 12 (n= 63) | -181.3 (198.25)
  Change from Baseline at Week 24 (n= 69) | -160.4 (185.45)
  Change from Baseline at Week 48 (n= 70) | -147.7 (191.63)

ADVERSE EVENTS:
Description: Only Treatment-Related Adverse Events were collected in this Post Marketing Surveillance Study.
Arm/Group | OZURDEX®
Serious Adverse Events (participants affected / at risk) | 1/99
Other Adverse Events (participants affected / at risk) | 26/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=99)
Endophthalmitis (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=99)
Ocular hypertension (Eye disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.